CLINICAL TRIAL: NCT03575884
Title: Fit 5 Kids Screen Time Reduction Curriculum for Latino Preschoolers: A RCT
Brief Title: Fit 5 Kids Screen Time Reduction Curriculum for Latino Preschoolers
Acronym: Fit5Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); Baylor College of Medicine (Other); USDA/ARS Children's Nutrition Research Center (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jason Mendoza, MD, MPH, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Fit5Kids R01; R01DK113005 (NIH)
Record Dates: First submitted 2018-06-12; First posted 2018-07-03 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Childhood; Physical Activity; Nutrition
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screen Time Reduction Curriculum (Experimental): Fit5Kids curriculum, weekly parent newsletters, in-person (or by telephone) goal setting on their child's screen time, a lending library of resources (books, games, arts/crafts, etc), and text messages on screen time parenting practices.
  Interventions: Behavioral: Screen Time Reduction Curriculum
- Control (No Intervention): Students will be taught the standard preschool curriculum.

INTERVENTIONS:
Behavioral: Screen Time Reduction Curriculum — Fit5Kids classroom curriculum, weekly parent newsletters, in-person (or by telephone) goal setting on their child's screen time, a lending library of resources (books, games, arts/crafts, etc), and text messages on screen time parenting practices offered over 7-8 weeks in the Fall semester. The classroom component will be taught by bilingual (English/Spanish) research staff interventionists. Parent newsletters, goal setting, and text messages will be offered in English and Spanish per parent preference. There will also be two "booster" weeks of classroom activities, daily parent newsletters, goal setting, and daily text messages on screen time parenting practices offered during the booster weeks in the Spring semester. The lending library of resources for parents/children will be available throughout the entire school year.
  Other Names: Fit5Kids
  Arms: Screen Time Reduction Curriculum

SUMMARY:
Childhood obesity and metabolic risk are at record high levels in the US, and Latino children are at very high risk. This project will test an intervention called Fit 5 Kids, designed for Latino preschoolers to decrease their screen time in order to promote physical activity and healthy eating, and to prevent obesity. Ultimately, this line of research has the potential to provide an effective program to reduce risk of obesity for Latinos in the Head Start program and other preschool-based settings.

DETAILED DESCRIPTION:
Screen time is a major risk factor for childhood obesity and inadequate physical activity, both of which are determinants of type 2 diabetes (T2D), cardiovascular disease, and multiple cancers. Latinos are the largest and fastest growing minority in the US. Because US Latino children have more screen time and higher rates of obesity than their non-Latino White peers, interventions to reduce screen time adapted for Latino preschoolers are necessary to reduce health inequities related to obesity and T2D in the US. However, a systematic review reported no successful screen time reduction interventions among Latino preschoolers.

The investigative team's pilot study tested the culturally adapted Fit 5 Kids screen time reduction curriculum among Latino preschoolers in Head Start. This short term cluster randomized controlled trial (RCT) is the only successful screen time reduction program for Latino preschoolers, having significantly reduced screen time by over 25 minutes/day. The investigative team's culturally adapted, multi-level intervention consists of lessons taught by study staff directly to preschoolers during Head Start, a weekly parent newsletter, and parenting tips via text messages several times/week. The investigative team will use a social ecological model and consider multiple levels of influences for analyses: (1) individual-level influences, e.g., acculturation and social cognitive theory, (2) families, e.g., screen time parenting practices, (3) schools, and (4) macro-environmental influences, e.g., neighborhood disorder. Building on this pilot work, the investigative team proposes a long term, efficacy, cluster RCT of the culturally adapted Fit 5 Kids among Latino preschoolers in Head Start from three US settings: Seattle, Houston, and the Central Valley of Washington State. Among 280 Latino 3-5 year olds at 20 Head Start centers, the investigative team's Specific Aims (SA) and Hypotheses (H) include:

SA1) To conduct a cluster RCT of the culturally adapted Fit 5 Kids curriculum to evaluate its efficacy in reducing screen time and excessive weight gain over a school year (8-months) H1) Fit 5 Kids will decrease children's screen time, BMI z-scores and dietary energy intake, and increase fruit/vegetable intake, skin carotenoids, and moderate/vigorous physical activity (MVPA) compared to controls

SA2) To examine mediators and moderators associated with reducing Latino preschoolers' screen time H2) Parents' outcome expectations, self-efficacy, and TV parenting practices will mediate the relationship between Fit 5 Kids and changes to preschoolers' screen time H3) Depressive symptoms, stress, and social support will moderate changes to preschoolers' screen time

The proposed Fit 5 Kids RCT will confirm the pilot's promising results, and the larger sample will allow for mediation analyses to better understand mechanisms. This research will provide justification for a future community effectiveness trial with implementation by Head Start teachers, and the eventual widespread implementation of Fit 5 Kids in Head Start centers nationally.

ELIGIBILITY:
Inclusion Criteria:

* Latino children, 3-5 years old, enrolled from 1 of the 20 Head Start Centers.
* Preschoolers do not require a minimum amount of screen time or devices in their household to enroll in the study, because it is preventive and population-based.
* Parents must be able to complete forms in English or Spanish.

Exclusion Criteria:

* Any preschooler that is underweight or under medical supervision to gain weight.
* Only one preschooler per family may be enrolled, to avoid clustering of variables by family.
* Preschoolers may only enroll once in the study.
* Children <3 years and >5 years of age.
* Children whose parents do not identify them as Latino or Hispanic.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Mendoza, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Research Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center - Center for Community Health Promotion, Sunnyside, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited from Head Start centers in three different regions: 1) Central Valley of Washington 2) Seattle, Washington 3) Houston, Texas. Research staff recruited a total of N= 22 schools and N=201 parent-child dyads to participate in the study. But, children were the focus of the intervention study outcomes. We report results pertaining to the children only. Head Start organizations in the three regions found centers for recruitment and those centers assisted in publicizing the trial.
Pre-assignment Details: Prior to randomization at Time 1, all assessments and surveys measuring mediating, moderating and outcome variables as well as covariates were assessed immediately pre-intervention at Time 1.
  Prior to randomization, we enrolled and consented 215 participants. Of those 215, 14 did not complete baseline assessments and/or were lost to follow -- these 14 participants were not randomized.
  Following Time 1, randomization occurred on a unit (Head Start school) level.
Units Other Than Participants: Head Start centers
Period: Overall Study
Arm/Group | Screen Time Reduction Curriculum | Control
Started | 92; 11 Head Start centers (92 children and 92 parents) | 109; 11 Head Start centers (109 children and 109 parents)
Completed | 92; 11 Head Start centers (92 children and 92 parents) | 109; 11 Head Start centers (109 children and 109 parents)
Not Completed | 0; 0 Head Start centers | 0; 0 Head Start centers

BASELINE CHARACTERISTICS:
Population: This data represents 92 parent child dyads in the intervention arm, and 109 parent child dyads in the control arm.11 schools were randomized into the Control Arm, likewise 11 schools were randomized into the Intervention Arm.
Groups:
- Screen Time Reduction Curriculum Child: Fit5Kids curriculum, weekly parent newsletters, in-person (or by telephone) goal setting on their child's screen time, a lending library of resources (books, games, arts/crafts, etc), and text messages on screen time parenting practices.
  Screen Time Reduction Curriculum: Fit5Kids classroom curriculum, weekly parent newsletters, in-person (or by telephone) goal setting on their child's screen time, a lending library of resources (books, games, arts/crafts, etc), and text messages on screen time parenting practices offered over 7-8 weeks in the Fall semester. The classroom component will be taught by bilingual (English/Spanish) research staff interventionists. Parent newsletters, goal setting, and text messages will be offered in English and Spanish per parent preference. There will also be two "booster" weeks of classroom activities, daily parent newsletters, goal setting, and daily text messages on screen time parenting practices offered during the booster weeks in the Spring semester. The lending library of resources for parents/children will be available throughout the entire school year.
- Control Child: Students will be taught the standard preschool curriculum.
- Total: Total of all reporting groups
Arm/Group | Screen Time Reduction Curriculum Child | Control Child | Total
Number analyzed (Participants) | 184 | 218 | 402
Age, Continuous [Mean (Standard Deviation); unit: years]
  Child Age | 4.6 (0.72) | 4.77 (0.64) | 4.69 (0.68)
  Parent Age | 30.39 (7.09) | 33.35 (8.02) | 32.01 (7.71)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Data represents parent-child dyads. They have been reported as child and parent respectively.
  Participants
    Sex of Child: number analyzed (Participants) | 92 | 109 | 201
    Sex of Child: Female | 40 | 52 | 92
    Sex of Child: Male | 48 | 49 | 97
    Sex of Child: Missing | 4 | 8 | 12
    Sex of Parent: number analyzed (Participants) | 92 | 109 | 201
    Sex of Parent: Female | 84 | 93 | 177
    Sex of Parent: Male | 4 | 7 | 11
    Sex of Parent: Missing | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data represents parent-child dyads. They have been reported as child and parent respectively.
  Participants
    Child Ethnicity: number analyzed (Participants) | 92 | 109 | 201
    Child Ethnicity: Hispanic or Latino | 87 | 95 | 182
    Child Ethnicity: Not Hispanic or Latino | 0 | 3 | 3
    Child Ethnicity: Unknown or Not Reported | 5 | 11 | 16
    Parent Ethnicity: number analyzed (Participants) | 92 | 109 | 201
    Parent Ethnicity: Hispanic or Latino | 86 | 97 | 183
    Parent Ethnicity: Not Hispanic or Latino | 2 | 2 | 4
    Parent Ethnicity: Unknown or Not Reported | 4 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data represents parent-child dyads. They have been reported as child and parent respectively.
  Participants
    Child Race: number analyzed (Participants) | 92 | 109 | 201
    Child Race: American Indian or Alaska Native | 0 | 0 | 0
    Child Race: Asian | 0 | 0 | 0
    Child Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child Race: Black or African American | 0 | 2 | 2
    Child Race: White | 69 | 82 | 151
    Child Race: More than one race | 2 | 4 | 6
    Child Race: Unknown or Not Reported | 21 | 21 | 42
    Parent Race: number analyzed (Participants) | 92 | 109 | 201
    Parent Race: American Indian or Alaska Native | 0 | 1 | 1
    Parent Race: Asian | 0 | 0 | 0
    Parent Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent Race: Black or African American | 0 | 1 | 1
    Parent Race: White | 69 | 80 | 149
    Parent Race: More than one race | 3 | 3 | 6
    Parent Race: Unknown or Not Reported | 20 | 24 | 44
Screen time [Mean (Standard Deviation); unit: minutes/day] — Unadjusted, children's screen time in minutes/day as measured by validated parent-reported screen time diaries
  minutes/day | 124.23 (79.38) | 127.28 (85.44) | 125.93 (82.57)

OUTCOME MEASURES:

1. Primary Outcome: Screen Time
Description: Screen Time Pre-intervention vs Post-intervention, measured by Screen Time Diary (7-day)
Time Frame: Week 1-2, Week 11-12, and Week 34-36
Measure: Mean (95% Confidence Interval); unit: minutes/day
Arm/Group | Screen Time Reduction Curriculum | Control
Number analyzed (Participants) | 92 | 109
minutes/day
  Week 1-2 (Time 1) | 122.6 [96.75 to 148.44] | 123.47 [99.58 to 147.35]
  Weeks 11-12 (Time 2) | 97.3 [70.74 to 123.86] | 129.34 [104.39 to 154.28]
  Weeks 34-36 (Time 3) | 122.85 [96.06 to 149.64] | 151.04 [125.46 to 176.62]
Statistical Analysis 1: Comparison: Screen Time Reduction Curriculum vs Control; Test type: Superiority; p < 0.05, Mixed Models Analysis; Study_arm timepoint interactions = -27.32, 95% CI 2-sided [-52.49 to -2.14]

2. Secondary Outcome: BMI Z-score
Description: Measured Height and Weight Pre-intervention vs Post-intervention. Body Mass Index (BMI) Z-score, is the child's calculated standard deviation from the CDC's population reference for child's sex and age. The formula is: Z-score = ((BMI / M)L - 1) / (L × S) where BMI is body mass index, M is median, L is the transformation for normality, and S is the coefficient of variations. A Z-score of 0 represents the mean for the CDC's reference population. Z-scores above the mean generally represent a worse outcome. A Z-score of 1.645 is the 95th percentile, which is considered the threshold for obesity.
  (info on the above can be found here: https://www.cdc.gov/growth-chart-training/hcp/computer-programs/sas.html)
Time Frame: Week 1-2, Week 11-12, and Week 34-36
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Screen Time Reduction Curriculum Child | Control Child
Number analyzed (Participants) | 92 | 109
score on a scale
  T1 | 1.04 [0.71 to 1.37] | 0.85 [0.48 to 1.22]
  T2 | 1.05 [.70 to 1.41] | 0.87 [0.49 to 1.25]
  T3 | 1.33 [.86 to 1.80] | 0.55 [0.09 to 1.02]

3. Secondary Outcome: Dietary Intake by Food Screener Data in Grams
Description: Dietary Intake Pre-intervention vs Post-intervention, measured by Block Kids Food Screener (more details below)
  Block Food Screeners for Ages 2-17 2007: These screeners are designed to assess children's intake by food group, with outcomes measured in number of servings. The version the investigative team will use for this study is about food eaten "last week." The focus of this tool is on intake of fruit and fruit juices, vegetables, potatoes (including French fries), whole grains, meat/poultry/fish, dairy, legumes, saturated fat, "added sugars" (in sweetened cereals, soft drinks, and sweets), glycemic load and glycemic index. A positive outcome would be to observe an increase in intake of fruit and vegetables, and reduced intake of saturated fats and added sugars.
Time Frame: Week 1-2, Week 11-12, and Week 34-36
Measure: Mean (95% Confidence Interval); unit: Grams
Arm/Group | Screen Time Reduction Curriculum Child | Control Child
Number analyzed (Participants) | 92 | 109
Grams
  T1 Saturated Fat in Grams | 13.93 [12.15 to 15.71] | 14.08 [12.50 to 15.66]
  T2 Saturated Fat in Grams | 13.99 [12.18 to 15.81] | 12.85 [11.20 to 14.50]
  T3 Saturated Fat in Grams | 15.16 [13.27 to 17.05] | 13.47 [11.73 to 15.20]
  T1 Sugar in Grams | 4.97 [4.17 to 5.76] | 4.72 [4.02 to 5.43]
  T2 Sugar in Grams | 4.89 [4.08 to 5.70] | 4.38 [3.65 to 5.12]
  T3 Sugar in Grams | 5.01 [4.17 to 5.85] | 4.94 [4.17 to 5.71]

4. Secondary Outcome: Fruit and Vegetable Intake and Skin Carotenoids
Description: Fruit and Vegetable Intake/Skin Carotenoid levels Pre-intervention vs Post-intervention, measured by Pharmanex BioPhotonic Scanner. Skin carotenoids are measured using Raman spectroscopy, which returned results in units of Raman counts from 0 to 70,000. Greater Raman counts indicate greater skin carotenoids and greater fruit/vegetable intake.
Time Frame: Week 1-2, Week 11-12, and Week 34-36
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Screen Time Reduction Curriculum Child | Control Child
Number analyzed (Participants) | 92 | 109
units on a scale
  Weeks 1-2 (Time 1) Skin Carotenoids | 26760.15 [16502.83 to 37017.48] | 26590.89 [16936.21 to 36245.57]
  Weeks 11-12 (Time 2) Skin Carotenoids | 36853.57 [26106.79 to 47600.36] | 28673.47 [18804.40 to 38542.54]
  Weeks 34-36 | 38017.93 [19313.15 to 56722.71] | 23030.60 [10777.72 to 35283.48]

5. Secondary Outcome: Physical Activity and Sedentary Behavior Time
Description: Physical Activity and Sedentary Behavior Time Pre-intervention vs Post-intervention, measured by ActiGraph Accelerometer GT3X+
Time Frame: Week 1-2, Week 11-12, and Week 34-36
Measure: Mean (95% Confidence Interval); unit: Minutes per Day
Arm/Group | Screen Time Reduction Curriculum Child | Control Child
Number analyzed (Participants) | 92 | 109
Minutes per Day
  T1 MVPA | 57.21 [47.57 to 66.86] | 66.15 [57.00 to 75.30]
  T2 MVPA | 58.66 [48.84 to 68.48] | 57.21 [47.81 to 66.61]
  T3 MVPA | 47.97 [37.55 to 58.40] | 49.53 [39.95 to 59.11]
  T1 Sedentary | 647 [534.96 to 760.78] | 719.67 [610.77 to 828.57]
  T2 Sedentary | 617.68 [503.79 to 731.58] | 649.30 [539.07 to 759.53]
  T3 Sedentary | 530.60 [413.01 to 648.20] | 625.02 [513.90 to 736.15]

6. Secondary Outcome: Dietary Intake by Food Screener Data in Cups
Description: as for outcome 3
Time Frame: Week 1-2, Week 11-12, and Week 34-36
Measure: Mean (95% Confidence Interval); unit: Cups
Arm/Group | Screen Time Reduction Curriculum Child | Control Child
Number analyzed (Participants) | 92 | 109
Cups
  T1 Fruit and Fruit Juice in Cups | 1.74 [1.46 to 2.02] | 1.57 [1.31 to 1.83]
  T2 Fruits and Fruit Juice in Cups | 1.62 [1.33 to 1.90] | 1.47 [1.20 to 1.73]
  T3 Fruits and Fruit Juice in Cups | 1.54 [1.25 to 1.83] | 1.54 [1.27 to 1.81]
  T1 Vegetables Without Potatoes in Cups | 0.64 [0.51 to 0.77] | 0.61 [0.49 to 0.73]
  T2 Vegetables Without Potatoes in Cups | 0.60 [0.47 to 0.74] | 0.52 [0.40 to 0.65]
  T3 Vegetables Without Potatoes in Cups | 0.60 [0.46 to 0.74] | 0.54 [0.42 to 0.67]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the academic year, i.e., over ~9 months for each cohort of randomized centers and parent child dyads. This data represents 92 parent child dyads in the intervention arm, and 109 parent child dyads in the control arm.
Arm/Group | Screen Time Reduction Curriculum | Control
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/109
Other Adverse Events (participants affected / at risk) | 0/92 | 0/109

LIMITATIONS AND CAVEATS:
The randomized controlled trial was conducted in part during the COVID-19 Pandemic and the results may have limited generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03575884/Prot_SAP_000.pdf